CLINICAL TRIAL: NCT02077998
Title: A Diagnostic Feasibility Trial of a [14C]Oxaliplatin Microdosing Assay for Prediction of Chemoresistance to Oxaliplatin Chemotherapy
Brief Title: Oxaliplatin in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#237; 457404 (Other: UC Davis); UCDCC#237 (Other: University of California, Davis); P30CA093373 (NIH); NCI-2013-01747 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (carbon C 14 oxaliplatin and oxaliplatin) (Experimental): PHASE 0: Patients receive carbon C 14 oxaliplatin IV over 2 minutes on day 1.
  PHASE II: Patients receive oxaliplatin IV over 2 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: carbon C 14 oxaliplatin; Drug: oxaliplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: carbon C 14 oxaliplatin — Given IV
  Other Names: [14C] oxaliplatin
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase 0/II trial studies the effect of carbon C 14 oxaliplatin in tumor tissue and blood and the side effects and how well oxaliplatin works in treating patients with metastatic breast cancer. DNA analysis of tumor tissue and blood samples from patients receiving carbon C 14 oxaliplatin may help doctors predict how well patients will respond to treatment with oxaliplatin. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To detect the levels of oxaliplatin-deoxyribonucleic acid (DNA) adducts induced by oxaliplatin microdosing in tumor tissue and peripheral blood mononuclear cells (PBMC), and correlate the results with patient response to oxaliplatin-based chemotherapy.

SECONDARY OBJECTIVES:

I. Evaluate the efficacy of single agent oxaliplatin treatment (130mg/m^2, 2 hr intravenously [IV] day 1; every 3 weeks) in pre-treated, metastatic breast cancer patients.

II. Evaluate the toxicity of oxaliplatin microdose and chemotherapy treatment in this patient population.

III. Determine the pharmacokinetic (PK) parameters of oxaliplatin microdosing and correlate with the PK parameters of therapeutic oxaliplatin.

IV. Determine whether the pharmacokinetics of oxaliplatin microdosing affects oxaliplatin-induced DNA damage and, therefore, patient response to chemotherapy.

V. Detect repair of DNA adducts in PBMC and correlate with patient response to oxaliplatin-based chemotherapy.

VI. Correlate the adduct and patient response data to DNA repair genes, such as excision repair cross-complementing (ERCC)1 levels as measured by reverse transcriptase-polymerase chain reaction (RT-PCR).

OUTLINE:

PHASE 0: Patients receive carbon C 14 oxaliplatin IV over 2 minutes on day 1.

PHASE II: Patients receive oxaliplatin IV over 2 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have metastatic breast cancer that can be biopsied or resected around 48 hours after dosing with one microdose of [14C]oxaliplatin (carbon C 14 oxaliplatin)
* Prior radiation or surgery is allowed, but should be finished at least 2 weeks prior to study enrollment; if a participant has prior radiation therapy, at least one measurable lesion outside of the radiation field should be available for the evaluation of response to chemotherapy
* Patients with metastatic breast cancer for which no standard therapy exists will be recruited for this study; more specifically, for patients with hormone receptor positive/human epidermal growth factor receptor 2 (Her2) negative disease, this includes previous therapy with tamoxifen or an aromatase inhibitor and one line of chemotherapy in the metastatic setting; for patients with Her2 positive disease, this includes 2 lines of Her2 directed therapy in the metastatic setting; and for patients with triple negative disease, this includes one line of chemotherapy in the metastatic setting; once we have identified the dose of [14C]oxaliplatin, we will only recruit triple negative breast cancer patients that progressed after one line of chemotherapy in the metastatic setting
* Any number of prior therapies other than oxaliplatin is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status equal to or less than 2 (Karnofsky equal to or greater than 50%)
* Life expectancy of at least 3 months
* Absolute neutrophil count greater than or equal to 1,500/microL
* Platelets greater than or equal to 100,000/microL
* Total bilirubin less than 1.5 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) less than or equal to 2.5 X ULN
* Creatinine less than 1.5 X ULN
* No pre-existing sensory neuropathy > grade 1
* Women of child bearing potential must not be pregnant; a pre-study pregnancy test must be negative
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 30 days after study participation
* Men must agree to use adequate contraception (barrier method or abstinence) prior to study entry and for 30 days after study participation
* Ability to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Patients must not receive concomitant radiation with chemotherapy if they do not have any measurable lesions outside of the radiation field
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Participants who are pregnant or nursing
* Participants who are allergic to platinum agent
* Participants who have more than grade 1 peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Threshold at which oxaliplatin-DNA adducts predict response to therapy | Up to 6 months post-treatment
  The concentration of oxaliplatin-DNA adducts induced will be characterized using descriptive statistics (graphical summaries, mean, standard deviation [SD], box plots) in PBMC and tumor for responders and non-responders to chemotherapy. The mean level of oxaliplatin-DNA adducts will be compared in responders to chemotherapy to that of non-responders using a 2-sample t-test at the 0.05 level (2-sided). The Youden index will be used to estimate and compute a 95% confidence interval for the optimal cut-point in oxaliplatin-DNA adduct levels to differentiate between responders and non-responders.

SECONDARY OUTCOMES:
Response rate assessed using Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 6 months post-treatment
  Will be analyzed primarily with respect to their association with level of oxaliplatin-DNA adducts. The distribution of clinical endpoints, including toxicity, will be summarized using frequencies for categorical data and Kaplan-Meier curves for survival data.
Progression-free survival | From the date of enrollment to the date of first objective evidence of radiographic progression (soft tissue or bone lesion) or date of death due to any cause, whichever occurs first, assessed up to 6 months post-treatment
  Will be analyzed primarily with respect to their association with level of oxaliplatin-DNA adducts. The distribution of clinical endpoints, including toxicity, will be summarized using frequencies for categorical data and Kaplan-Meier curves for survival data.
Overall survival | From the first treatment to death or to the last treatment follow-up, assessed up to 6 months post-treatment
  Will be analyzed primarily with respect to their association with level of oxaliplatin-DNA adducts. The distribution of clinical endpoints, including toxicity, will be summarized using frequencies for categorical data and Kaplan-Meier curves for survival data.
Overall toxicity from both the carbon C 14 oxaliplatin microdose and the full dose oxaliplatin chemotherapy evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days post-treatment
  Will be analyzed primarily with respect to their association with level of oxaliplatin-DNA adducts. The distribution of clinical endpoints, including toxicity, will be summarized using frequencies for categorical data and Kaplan-Meier curves for survival data. Safety will be assessed through summaries of adverse events, the frequency of treatment discontinuations due to adverse events, and laboratory evaluations. Descriptive statistics will be used rather than inferential statistics.
PK parameters including maximum concentration (Cmax), half-life (t1/2), and area under the curve (AUC) from both micro- and therapeutic- dosing in the same patients | Pre-dose; 5, 15, and 30 minutes; and 2, 4, 8, 24, and 48 hours
  PK parameters from microdosing will be correlated with parameters from therapeutic dosing. Descriptive summaries (scatterplots, tables, mean, SD, correlation coefficient) of the relationship between the two sets of parameters will be presented.
Levels of oxaliplatin-DNA adducts in tumor and PBMC | Up to 48 hours
  Responders and non-responders will be compared using two-sample t-tests; if the half-lives are not normally distributed, Wilcoxon rank-sum tests will be used. The effect of half-life on progression-free survival will be explored using Cox proportional hazards models. Similar analyses will be performed for other PK parameters.
Repair of oxaliplatin-DNA monoadducts in PBMCs | Up to 48 hours
  Will be characterized using descriptive statistics (graphical summaries, mean, SD, box plots).
Messenger ribonucleic acid (mRNA) expression levels of ERCC1 | Up to 48 hours
  Descriptive statistics, such as graphical summaries, mean, SD, box plots will be used for responders and non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Xian Pan, Principal Investigator — UC Davis Cancer Center
Locations (1):
- UC Davis Comprehensive Cancer Center, Sacramento, California, United States